CLINICAL TRIAL: NCT04922437
Title: Site of Implantation of Continent Catheterizable Channel : Native Bladder or Enterocystoplasty ? Comparison in 106 Patients
Brief Title: Implantation of Continent Catheterizable Channel : Native Bladder or Enterocystoplasty ?
Acronym: ICODE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pierre LECOANET, Doctor, Central Hospital, Nancy, France
Other Study IDs: 2020PI311
Record Dates: First submitted 2021-05-24; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Neurogenic Bladder; Continent Cutaneous Urinary Diversion; Mitrofanoff
Keywords: native bladder; enterocystoplasty; continent catheterizable channel; neurogenic bladder
MeSH Terms: conditions — Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Enterocystoplasty (EC): Patients who had an implantation of the catheterizable continent channel by seromuscular plicature on the anterior wall of the bladder augmentation.
  Interventions: Procedure: Enterocystoplasty implantation
- Detrusor (D): Patients who had an implantation of the catheterizable continent channel in the detruosr of their native bladder (Lich-Gregoir or Cohen).
  Interventions: Procedure: Native bladder implantation

INTERVENTIONS:
Procedure: Native bladder implantation — Continent catheterizable channel implanted in the detrusor of the native bladder
  Groups: Detrusor (D)
Procedure: Enterocystoplasty implantation — Continent catheterizable channel implanted by seromuscular plicature on the front wall of the bladder augmentation
  Groups: Enterocystoplasty (EC)

SUMMARY:
PURPOSE. To compare the results between two sites of implantation of the continent catheterizable channel (CCC): native bladder or enterocystoplasty.

METHODS. Retrospective monocentric study of pediatrics and adult patients who underwent a continent cystostomy between 1991 and 2020 with a continent catheterizable channel implanted in the native bladder's detrusor (D group) or the enterocystoplasty (EC group).

DETAILED DESCRIPTION:
This is a monocentric and retrospective study involving adult and pediatric population who underwent the creation of a CCC between June 1991 and January 2020. Two different surgical techniques were performed: on the first hand, the implantation of the channel in the native bladder's detrusor (D group), on the other hand the implantation of the channel by seromuscular plicature on the anterior wall of the enterocystoplasty (EC group).

The CCC were made from the appendix, an ileal or sigmoid segment, an ureter or a skin flap. Bladder augmentation and cervicoplasty (Kropp, Kurzrock, Young-Dees, artificial urinary sphincter, sling suspension of the bladder neck, closure of the bladder neck) were frequently associated.

The following informations were obtained in all included patients by charts reviews: age at surgery, gender, main underlying pathology, details of operative reports with the type of channel, bladder augmentation and/or associated cervicoplasty, early postoperative complications, complications appearing during the follow up period and the requirement of surgical or non-surgical revision, finally the channel continence at the last follow up.

ELIGIBILITY:
Inclusion Criteria:

* Adult and pediatric patients who underwent a surgery for creation of a continent catheterizable channel
* Between 1991 and 2020
* In the pediatric surgery or urology department at Nancy University Hospital

Exclusion Criteria:

* Ghoneim technique used for implantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric population recruited in the pediatric surgery and urology departments of Nancy University Hospital. Patients with congenital or acquired neurological bladder or malformative uropathies.
  Surgery performed between 1991 and 2020, followed in the long term in iterative consultation or in hospitalization for evaluation of continence and postoperative complications with or without surgical revision
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of the long term continence between the two groups | 1 year
  Continence of the channel at last followup : as being strictly dry day and night between clean intermittent catheterizations (CIC). Patients requirring at leat one pad for leaking and also those with leaks wetting their clothes were considered incontinent as well as those whose interval between CIC was strictly less than 3 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Lecoanet, Principal Investigator — CHRU Nancy
Locations (1):
- Pierre Lecoanet, Vandœuvre-lès-Nancy, France